CLINICAL TRIAL: NCT06268249
Title: Ulinastatin Improves Post-Cardiac Surgery Cognitive Dysfunction by Inhibiting Glycocalyx Degradation: An Observational Study
Brief Title: Ulinastatin Improves Post-Cardiac Surgery Cognitive Dysfunction
Status: Completed | Type: Observational
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20231224
Record Dates: First submitted 2024-02-04; First posted 2024-02-20 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium
Keywords: POCD - Postoperative Cognitive Dysfunction; POD-Postoperative Delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium | interventions — urinastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ulinastatin — Ulinastatin was pumped continuously during the operation

SUMMARY:
The study comprised two primary components: a retrospective analysis of clinical big data and a conventional prospective cohort study involving patients undergoing cardiac surgery. The objectives were: 1. To assess the preventive effect of ursodeoxycholic acid on post-cardiac surgery cognitive dysfunction over an eight-year period. 2. To analyze preoperative and postoperative 24-hour plasma samples from prior studies to quantify the levels of glycocalyx and its associated regulatory factors. 3. To evaluate the clinical association between the measured parameters and patient outcomes.

DETAILED DESCRIPTION:
1. Baseline Period Visit 1 (within 24 hours before surgery)

   Sign informed consent Check inclusion/exclusion criteria Demographic data (sex, age, occupation, etc.) Past medical history (stroke, hypertension, diabetes, dyslipidemia, coronary heart disease, diabetes, etc.) and medication history in the past 3 months Vital signs (temperature, pulse, respiration, blood pressure) Preoperative ECG Preoperative echocardiography Laboratory tests (blood routine, blood glucose, blood lipids, liver and kidney function, myocardial enzymes, blood electrolytes, coagulation function) Concomitant therapy Adverse events
2. Intraoperative cardiopulmonary bypass

   Record vital signs and various physiological indicators in the operating room. Routinely perform central venous puncture to establish venous access and monitor central venous pressure, and radial artery puncture to monitor invasive arterial pressure.

   After general anesthesia and endotracheal intubation, routine blood chemistry and arterial blood gas analysis were performed.

   After collecting the above blood samples for testing, the remaining blood was centrifuged, and the plasma was frozen at -80°C for subsequent testing (levels of CRP, IL-6, IL-10, TNF-α, TK/B1R/MMP3, Hyaluronic acid, etc.).

   Operation time Vital signs (temperature, pulse, respiration, blood pressure) Routine blood chemistry and arterial blood gas analysis Document vasoactive drug use
3. 24 hours, 72 hours, 7 days after surgery

   Vital signs (temperature, pulse, respiration, blood pressure) Bedside echocardiography Laboratory tests (blood routine, blood sugar, blood lipids, liver and kidney function, myocardial enzymes, coagulation function, etc.) After collecting the above blood samples for testing, the remaining blood is centrifuged, and the plasma is frozen at -80°C for later testing (levels of glycocalyx) POCD Document treatment regimen (including vasoactive drug use, etc.)
4. Follow-up period

CCU time and total hospital stay 28-day survival status The survival status of the patients was followed up, and the date of death and the cause of death should be recorded in the patients who died.

Research Evaluation Analyze the clinical correlation between glycocalyx and its related indicators and postoperative cognitive dysfunction after cardiac surgery.

Patient Completion/Withdrawal from Study Finish All evaluation data of the patients 28 days after the operation were completely collected and considered as completed cases.

Inclusion criteria:

Voluntary participation in the study; Age ≥ 18 years and ≤ 80 years; Patients undergoing heart surgery: (heart valve replacement surgery with CPB,coronary artery bypass grafting, Morrow procedure, aortic dissection surgery).

Exclusion criteria:

Recipients of solid organ or bone marrow transplants; Patients with autoimmune diseases, tumors, or who have received high-dose steroids or immunosuppressive therapy within the past 2 months; Deemed unsuitable for participation in this study by the researchers. Primary outcome: Postoperative Delirium, postoperative cognitive dysfunction. Objective: Analyze the correlation between polysaccharide coating and cardiac surgery-related indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the study;
2. Age ≥ 18 years and ≤ 80 years;
3. Patients undergoing heart surgery: (coronary artery bypass grafting, heart valve replacement surgery, Morrow procedure, aortic dissection surgery).

Exclusion Criteria:

1. Patients experiencing adverse events during the surgery;
2. Recipients of solid organ or bone marrow transplants;
3. Patients with autoimmune diseases, tumors, or who have received high-dose steroids or immunosuppressive therapy within the past 2 months;
4. Deemed unsuitable for participation in this study by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing heart surgery: (coronary artery bypass grafting, heart valve replacement surgery, Morrow procedure, aortic dissection surgery).
Sampling Method: Non-Probability Sample
Enrollment: 7065 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
POCD - Postoperative Cognitive Dysfunction | 24 hours
  Mini-Mental State Examination（MMSE）
POD-postoperative delirium | 7 days
  Confusion Assessment Method for the ICU (CAM-ICU)

SECONDARY OUTCOMES:
Survival time | 28 days
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ran X, Xu T, Liu J, Yang S, Luo F, Wu R, Tan J, Ruan H, Zhang Q. Ulinastatin treatment mitigates glycocalyx degradation and associated with lower postoperative delirium risk in patients undergoing cardiac surgery: a multicentre observational study. Crit Care. 2025 Jan 29;29(1):52. doi: 10.1186/s13054-025-05296-9. PMID 39881341